CLINICAL TRIAL: NCT04568616
Title: Phase II Study of Neoadjuvant ArOMatase Inhibitor Therapy for ER+ Breast Cancer (NAOMI)
Acronym: NAOMI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Mary D Chamberlin, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D20148; NCI-2022-02378 (Other: NCI ID)
Record Dates: First submitted 2020-09-22; First posted 2020-09-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; ER Positive Breast Cancer
Keywords: Letrozole; Aromatase Inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Intervention Model Description: Patients receive letrozole orally (PO) once daily (QD) for 4-16 weeks up to the day of surgery in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery. After surgery, a subset of patients start a hormone therapy (letrozole, anastrozole, or tamoxifen) and remain in the study for up to 3.5 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Letrozole 2.5mg tablet administered once daily for 4 to ~12 weeks (window of + 4 weeks for surgical scheduling flexibility) final dose taken the day of surgery.
  Interventions: Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: Letrozole 2.5mg — Aromatase Inhibitor
  Other Names: Femara

SUMMARY:
This is a single-arm, open-label study testing the effects of neoadjuvant therapy with the aromatase inhibitor letrozole in post-menopausal women with Stage I-III ER+, HER2- breast cancer. Eligible subjects will be treated with letrozole therapy for 4 to 24 weeks prior to surgical resection of the tumor. Tumor specimens obtained at baseline (diagnostic biopsy) and at surgery (surgical specimen) will be compared using molecular analyses. A subset of subjects will be asked to provide an optional research tumor biopsy prior to treatment for molecular analysis. Subjects will be evaluated for treatment adherence and provide feedback via survey questionnaires to identify potential causes of non-adherence.

DETAILED DESCRIPTION:
Approximately 70% of breast cancers express estrogen receptor alpha (ER), which is activated by estrogens and typically drives cancer cell growth. Adjuvant therapy with anti-estrogens such as tamoxifen and aromatase inhibitors (AIs) is commonly used to inhibit ER to prevent cancer (re)growth after early-stage breast tumors are surgically removed. However, ~33% of such patients (~300,000 new cases per year worldwide) will eventually develop anti-estrogen-resistant breast cancer that is metastatic or locally advanced; at this stage, the disease is almost never cured using available therapies and is uniformly fatal. Therefore, more effective treatment early in the course of disease (i.e., in the adjuvant setting, shortly after surgical removal of a tumor) has huge potential to prevent cancer regrowth. Most often, ER+ breast cancers re-emerge in the years after the end of the standard five-year anti-estrogen treatment regimen (called 'late recurrence'). Recent data indicate that continued anti-estrogen therapy in patients who remain "disease-free" after five years of anti-estrogen therapy modestly prevents cancer recurrence. However, tumor cells are detectable in bone marrow of patients who are "disease-free." Thus, antiestrogen therapy in "disease-free" patients likely suppresses the growth of undetectable tumor cells, keeping them in a "clinically dormant" state (i.e., undetectable by standard clinical methods). Little is known about how such dormant cancer cells survive. This clinical study will help identify the signaling pathways essential for the survival of clinically dormant ER+ breast cancer cells to enable the development of more effective therapies to eradicate such cells and prevent cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic documentation of invasive breast cancer by core needle or incisional biopsy. Subjects without excess baseline tumor tissue are eligible and evaluable for Primary Objective #2 (re: adherence). Excess baseline biopsy tumor tissue sufficient to make ten 5- micron sections must be available for research use for a subject to be evaluable for Primary Objective #1 (re: molecular analyses).
2. The invasive cancer must be estrogen receptor alpha (ER)-positive, with ER staining present in greater than 50% of invasive cancer cells by IHC.
3. The invasive cancer must be HER2-negative (IHC 0-1+, or with a FISH ratio of <1.8 if IHC is 2+ or if IHC has not been done).
4. Clinical Stage I-III invasive breast cancer with the intent to treat with surgical resection of the primary tumor. Baseline tumor must be ≥0.5 cm. For the optional research biopsy (from 5 subjects), tumor must be

   ≥1 cm.
5. Patients with multicentric or bilateral disease are eligible if the subject is a candidate for clinically indicated neoadjuvant endocrine therapy. Samples from all available tumors are requested for research purposes.
6. Women over 18 years of age, for whom (A) neoadjuvant treatment with an aromatase inhibitor would be clinically indicated, and (B) adjuvant treatment with one of the following would be clinically indicated: tamoxifen; anastrozole; letrozole. Women must be postmenopausal, defined as last menstrual period >2 years prior to registration, or >1 yearer prior to registration with FSH and estradiol in post-menopausal range.
7. Patients must meet the following clinical laboratory criteria:

   * Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet count ≥ 75,000/mm3.
   * Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
8. Ability to give informed consent.

Exclusion Criteria:

1. Prior endocrine therapy for any histologically-confirmed cancer or prevention of breast cancer in the last 10 years is not allowed.
2. Any other neoadjuvant therapy for breast cancer. Bisphosphonate or denosumab treatment for metabolic bone issues are allowed.
3. Women who are pregnant or lactating.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2029-08-13 (Estimated)

PRIMARY OUTCOMES:
Change in Tumor CPT1-alpha levels | Baseline to 4-12 Weeks
  Determine whether residual cancer cells exhibit upregulation of the fatty acid transport CPT1-alpha (compared to baseline) following neoadjuvant endocrine therapy in patients with ER+ breast cancer.
Determine subject adherence to endocrine therapy as measured via urine analysis | Before surgery (within 14 days before surgery, or on day of surgery); approximately 1 year after surgery; and approximately 3 years after surgery
  Urine analysis for drug metabolites will be used to determine subject adherence to endocrine therapy at three time points. (Protocol section 6.16.e) The outcome measure is percent of participants with adherence vs non-adherence as measured by urine samples tested for metabolites of adjuvant endocrine agents: tamoxifen, letrozole, anastrozole or exemestane. Urine tests will be recorded as positive or negative. Positive urine test = adherence.
Treatment Satisfaction Questionnaire for Medication (TSQM) side effects score | Before surgery (approximately 4-24 weeks after the start of letrozole treatment), 1 year after surgery, and 3 years after surgery
  The Treatment Satisfaction Questionnaire for Medication (TSQM) v1.4 assesses subjects' satisfaction with their breast cancer medication over the past 2-3 weeks, or since last use. A modified 12-item questionnaire will address 4 domains: effectiveness (Item 1), side effects (Items 2-6), convenience (Items 7-9), and global satisfaction (Items 10-12). Item 2 (experience of side effects; yes/no) will be evaluated independently. Subjects will be dichotomized at the median score for analysis.

SECONDARY OUTCOMES:
Longest dimension(s) of primary tumor(s) pre- and post-treatment | Baseline and after approximately 4 to 24 weeks of treatment
  The longest dimension(s) of the primary tumor(s) will be measured from radiological images acquired as per standard of care before neoadjuvant letrozole treatment, and after neoadjuvant letrozole treatment (prior to surgery). If multiple primary tumors are detected, the sum of the longest diameters will be used to provide a single measurement at each time point for each subject. Pre- and post-treatment tumor lengths will be compared.
Altered mitochondrial and fatty acid metabolism in surgical tissue specimen as compared to baseline tissue specimen. | Baseline and at surgery (after approximately 4 to 24 weeks of treatment)
  Sections of baseline and post-neoadjuvant therapy tumor tissue specimens will be immunofluorescently stained using antibodies against TOM-20, ACC, FASN, CD36, and perilipin. Mitochondrial number and length (per cancer cell) will be measured using Halo software to determine whether neoadjuvant therapy cancer cells exhibit increased mitochondrial content compared to baseline cancer cells. Other markers will be scored by Histoscoring. Correlations between A) the duration of neoadjuvant letrozole, and B) expression of metabolic markers (CPT1-alpha, TOM-20, FASN, CD36, perilin) will be determined.
Brief Pain Inventory (BPI) scores | Baseline (within 28 days prior to start of letrozole), Before surgery (approximately 4-24 weeks after the start of letrozole treatment), 1 year after surgery, and 3 years after surgery
  The Brief Pain Inventory (BPI) asks subjects to rate pain (modified to also include stiffness) over the prior week and the degree to which it interferes with activities on a 0 to 10 scale, where higher scores indicate more pain or interference. We will examine items reflecting worst pain, least pain, average pain, pain right now, and pain interference. Pain interference will be calculated as the mean score across 7 items (in Question 9). Subjects will be dichotomized at the median score using each of the above metrics, and rates of non-adherence will be calculated for subjects below vs. above the median.
Functional Assessment of Cancer Therapy- Endocrine Symptoms (FACT-ES) scores | Baseline (within 28 days prior to start of letrozole), Before surgery (approximately 4-24 weeks after the start of letrozole treatment), 1 year after surgery, and 3 years after surgery
  The Functional Assessment of Cancer Therapy-Endocrine Symptoms (FACT-ES) contains (A) the Functional Assessment of Cancer Therapy- General (FACT-G) to measure physical, social, family, emotional, and functional well-being through 4 subscales, and (B) a fifth 18-item subscale to measure endocrine-related symptoms. In FACT-G, 6-7 items are queried in each subscale. FACT scales have 5 response levels ("not at all" to "very much"), where higher scores reflect increased wellness. The sum of item scores in each subscale will be calculated, multiplied by the number of items in the subscale, and divided by the number of items answered to derive a subscale score for each subject. The sum of subscale scores will yield the total FACT-G and FACT-ES score for each subject. Subjects will be dichotomized at the median scores for analysis.
Beliefs about Medication Questionnaire (BMQ) score | Baseline (within 28 days prior to start of letrozole), Before surgery (approximately 4-24 weeks after the start of letrozole treatment), 1 year after surgery, and 3 years after surgery
  The Beliefs about Medication Questionnaire (BMQ) assesses patients' beliefs about their prescribed medication. BMQ items were adapted to reflect medication prescribed for cancer. Subjects will indicate their degree of agreement with each statement on a 5-point Likert scale ("strongly disagree" to "strongly agree"). The sum of scores for all items will be calculated for each subject. Subjects will be dichotomized at the median score for analysis.
Treatment Satisfaction Questionnaire for Medication (TSQM) total and domain scores for effectiveness, convenience, global satisfaction, and experience of side effects | Before surgery (approximately 4-24 weeks after the start of letrozole treatment), 1 year after surgery, and 3 years after surgery
  1. Change in Treatment Satisfaction Questionnaire for Medication (TSQM) total
  2. Change in Treatment Satisfaction Questionnaire for Medication (TSQM) for effectiveness
  3. Change in Treatment Satisfaction Questionnaire for Medication (TSQM) for convenience
  4. Change in Treatment Satisfaction Questionnaire for Medication (TSQM) for global satisfaction
Endocrine Therapy adherence pre and post surgery. | Baseline to 4 -12 weeks
  Determine the proportion of subjects who receive ≥1 wk of neoadjuvant endocrine therapy and remain adherent with prescribed adjuvant endocrine therapy at 1 and 3 years post surgery.
Proportion of subjects who experience Clinical Response | 4 to12 Weeks
  Determine the proportion of subjects who experience clinical response, defined as a ≥50% decrease in the longest dimension of the primary tumor(s) measured from the start of treatment to right before surgery.

OTHER OUTCOMES:
Changes in residual cancer fatty acid. | Baseline to 4 -12 weeks
  Compare values of CPT1-alpha histoscores in pre and post neoadjuvant endocrine therapy samples to show the number of samples with residual disease that exhibit upregulation of the fatty acid transporter CPT1-alpha compared to pre-treatment samples.
Changes in tumor cell type | Baseline to 4 -12 weeks
  Using fresh tumor tissue at baseline, tumor cell type proportions before and after neoadjuvant endocrine therapy will be measured per 10X Genomics manufacturer's protocol. Data will be bioinformatically analyzed using dimensionality reduction with t-distributed stochastic neighbor embedding (t-SNE) to visualize data in two dimensions and measure:
  1. Percent of each cell type before and after neoadjuvant endocrine therapy
  2. Change in cell type proportions via t-SNE
Relationship between duration of endocrine therapy and changes in tumor markers. | Baseline to 4 -12 weeks
  Determine whether duration of neoadjuvant letrozole treatment is correlated with changes in markers of altered mitochondrial and fatty acid metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Mary D Chamberlin, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- United States (2):
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire